CLINICAL TRIAL: NCT04589013
Title: Prediction of Response to Treatment With Immunotherapy + Chemotherapy in Non-Small Cell Lung Cancer
Acronym: PRINCE
Status: Completed | Type: Observational
Sponsor: University Hospital, Lille (Other)
Responsible Party: Sponsor
Other Study IDs: 2019_06; 2019-A03156-51 (Other: ID-RCB number,ANSM)
Record Dates: First submitted 2020-10-08; First posted 2020-10-19 (Actual); Last update posted 2025-12-23 (Actual); Status verified 2025-12

CONDITIONS: Non-small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study seeks to evaluate a multiparametric test including 6 immunohistochemical markers (PD-L1, CD8, FoxP3, PD1, CD163, CD15) to predict the cumulative incidence of death or progression on treatment with pembrolizumab+first line chemotherapy in metastatic non-small cell lung cancer, regardless of the PD-L1 status and in the absence of ALK, ROS1 or EGFR alteration.

ELIGIBILITY:
Inclusion Criteria:

* 18 years at time of diagnosis
* Affiliation to a social insurance
* Obtaining the patient's non opposition
* Patients with non-small cell lung carcinoma, confirmed by anatomopathological, metastatic or locally advanced unresectable, not eligible for local curative treatment
* Cellular or tissue FFPE available
* Indication of treatment with pembrolizumab + first line chemotherapy in multidisciplinary consultation meeting
* No mutation of the EGFR gene, no rearrangement of ALK and ROS,
* At least one measurable tumor according to RECIST criteria

Exclusion Criteria:

* Tissue or cellular FFPE not available
* Systemic anti-neoplastic or immunotherapy previously received except neoadjuvant or adjuvant treatment completed 6 months or more

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients meeting the inclusion criteria will be selected in each of the centers (Lille CHU, Lille Centre Oscar Lambret, Valenciennes Clinique Teissier, Roubaix CH) by the onco-pneumologists and included in the study, after collecting the consent, at the start of treatment with pembrolizumab + chemotherapy in first line.
Sampling Method: Probability Sample
Enrollment: 106 (Actual)
Dates: Start 2020-11-19 (Actual); Primary Completion 2023-09-29 (Actual); Study Completion 2023-09-29 (Actual)

PRIMARY OUTCOMES:
The dependent variable will be the cumulative incidence of death or progression under immunotherapy + chemotherapy at 1 year. | At 1 year
  Progression will be evaluated by CT imaging every 12 weeks and then every 9 weeks according to RECIST 1.1.
  The independent variables will be the 6 immunohistochemical markers (PD-L1, CD8, FoxP3, PD1, CD163, CD15) evaluated prior to the first injection of pembrolizumab + chemotherapy from the diagnostic tissue material.

SECONDARY OUTCOMES:
Discrimination index (concordance index=C-statistics) of the multiparametric model and model including that of the PD-L1 test. | At 1 year
  Compare the discriminant power of the multiparametric model to that of the PD-L1 test alone.

CONTACTS AND LOCATIONS:
Overall Officials: Sarah Humez, Principal Investigator — University Hospital, Lille
Locations (4):
- France (4):
  - Clcc Oscar Lambret Lille, Lille
  - Hop Calmette Chu Lille, Lille
  - CH Victor Provot, Roubaix
  - Clinique Teissier, Valenciennes